CLINICAL TRIAL: NCT04350580
Title: Value of Early Treatment With Polyvalent Immunoglobulin in the Management of Acute Respiratory Distress Syndrome Associated With SARS-CoV-2 Infections
Brief Title: Polyvalent Immunoglobulin in COVID-19 Related ARds
Acronym: ICAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Groupe Hospitalier Universitaire Paris psychiatrie & neurosciences (Unknown); Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D20-P013; 2020-001570-30 (EudraCT Number)
Record Dates: First submitted 2020-04-08; First posted 2020-04-17 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Acute Respiratory Distress Syndrome; COVID-19
Keywords: acute respiratory distress syndrome; COVID-19; SARS-CoV-2; Immunoglobulin
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19 | interventions — Immunoglobulins, Intravenous; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The participant will be randomized to either the group of treatment with IVIG or the placebo group. Participants in the treatment group will receive infusions of polyvalent immunoglobulins for 4 consecutive days. Participants in the placebo group will receive an equivalent volume of sodium chloride 0.9% for the same duration.
Who Masked: Participant, Care Provider
Masking Description: The double blinding will be provided by the hospital pharmacy of each establishment with the help of opaque sleeves to mask the product packaging and should be returned to the pharmacy when empty.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention - IGIV (Experimental): Participants in the intervention group will receive a 2g/Kg infusion of human immunoglobulin which should be started before the 96th hours after the start of mechanical ventilation in 4 injections of 0.5 g/Kg over 4 consecutive days.
  Interventions: Drug: Human immunoglobulin
- Placebo (Placebo Comparator): Participants of the placebo group will receive an equivalent volume of sodium chloride 0.9% for the same duration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Human immunoglobulin — Human immunoglobulin 2g/kg over 4 days (0.5g/kg/d)
  Other Names: Clairyg
  Arms: Intervention - IGIV
Drug: Placebo — Sodium chloride 0.9% in the same volume and over the same time as the immunoglobulin
  Other Names: Sodium chloride 0.9%
  Arms: Placebo

SUMMARY:
As of 30/03/2020, 715600 people have been infected with COVID-19 worldwide and 35500 people died, essentially due to respiratory distress syndrome (ARDS) complicated in 25% of the with acute renal failure. No specific pharmacological treatment is available yet. The lung lesions are related to both the viral infection and to an intense inflammatory reaction. Because of it's action, as an immunomodulatory agent that can attenuate the inflammatory reaction and also strengthen the antiviral response, it is proposed to evaluate the effectiveness and safety of intravenous immunoglobulin administration (IGIV) in patients developing ARDS post-SARS-CoV2. IGIV modulates immunity, and this effect results in a decrease of pro-inflammatory activity, key factor in the ARDS related to the COVID-19. It should be noted that IGIV is part of the treatments in various diseases such as autoimmune and inflammatory diffuse interstitial lung diseases. In addition, they have been beneficial in the post-influenza ARDS but also have been in 3 cases of post-SARS-CoV2 ARDS. IGIV is a treatment option because it is well tolerated, especially concerning the kidney. These elements encourage a placebo-controlled trial testing the benefit of IGIV in ARDS post-SARS-CoV2.

DETAILED DESCRIPTION:
As of 30/03/2020, 715600 people have been infected with COVID-19 worldwide and 35 500 people have died, mainly from acute respiratory distress syndrome (ARDS) complicated in 25% of cases with acute renal failure. No specific pharmacological treatment is available yet. Pulmonary lesions in these patients are related to both viral infection and an inflammatory reaction. Patients admitted to intensive care have an important inflammatory response and increased plasma concentrations of IL2, IL7, IL10, GCSF, IP10, MCP1, MIP1A, and TNFα.

In the blood, the number of peripheral CD4 and CD8 T cells appears to be significantly reduced, while their status is hyperactivated. This is evidenced by immunoreactive cytometrics for HLA-DR (CD4 3-47%) and CD38 (CD8 39-4%) or by an increase in the proportion of highly pro-inflammatory Th 17 CCR6+ lymphocytes. In addition, CD8 T cells would exhibit a highly cytotoxic profile characterized by high concentrations of cytotoxic granules, perforin+, granulysin+ or double positive, suggesting associated complement activation. Because of their immunomodulatory action, which can attenuate the inflammatory response; and also strengthen the anti-viral defence, it is proposed to evaluate the efficacy and safety of intravenous immunoglobulin (IGIV) administration in patients developing post-SARS-CoV2 ARDS.

IGIV modifies cell function of dendritic cells, cytokine and chemokine networks and T-lymphocytes, resulting in the proliferation of regulatory T cells to regulate the activity of T lymphocytes CD4 or CD8. The action of IGIV induces an activation more particularly of lymphocytes T regulators that could modulate the effects of the lymphocyte populations described in the study by Xu et al during COVID-19. In addition, IGIV modulate humoral acquired immunity, through their effect on the idiotypic network and antibody production. They also act on innate immunity, through antigen neutralization and modulation of phagocytic cells. These effects result in a decrease in the production of pro-inflammatory cytokines and complement activation, key factors in post-SARS-CoV2 ARDS.

IGIV is part of the treatment for a variety of autoimmune and inflammatory diseases. The standard IGIV as well as polyclonal IGIV significantly reduced mortality in patients with septic shock and in Kawasaki disease, which is post-viral vasculitis of the child. In addition, they would not only be beneficial in post-influenza ARDS, but also would also in 3 cases of post-SARS-CoV2 ARDS. IVIG is a treatment option because it is well tolerated, especially regarding renal function.

These factors are encouraging to quickly conduct a multicentre randomized placebo-controlled trial testing the benefit of IGIV in post-SARS-CoV2 ARDS.

We hypothesize that the number of days without invasive mechanical ventilation (IMV) is 10 days in the placebo group and 15 days in the experimental group with a standard deviation of 6 days, considering a mortality of 50% and 40% in the placebo and experimental groups respectively (26, 27). The number of days without IMV in the placebo group is (50% x 10 D) + (50% x 0 D) or 5 D on average, and following the same calculation for the experimental group of (60% x 15 D) + (40% x 0 D) or 9 D.

Therefore, a mean value of 5 days without ventilation in the placebo group versus 9 in the experimental group is assumed, and the 6-day standard deviation is assumed to be stable. Given the uncertainty regarding the assumption of normality of distributions, the non-parametric Wilcoxon-Mann-Whitney test (U-test) was used for the estimation of the sample size. Considering a bilateral alpha risk of 5% and a power of 90% and an effect size of 0.6, the number of subjects to be included is 138 patients, 69 in each arm.

The primary and secondary analyses will be stratified by age categories, sex and other clinically relevant factors (comorbidities). Demographic characteristics and parameters identified at enrolment will be summarized using descriptive statistical methods.

Demographic summaries will include gender, race/ethnicity, and age. For demographic and categorical background characteristics, a Cochran-Mantel-Haenszel test will be used to compare treatment groups. For continuous demographic and baseline characteristics, a Wilcoxon test will be used to compare treatment groups.

The number of days without mechanical ventilation will be presented as a mean with standard deviation. The groups will be analyzed in terms of intention to treat and the difference between the two groups will be analyzed by a non-parametric test of comparison of means, stratified for the primary endpoint. The point estimate of the difference between treatments and the associated 95% confidence interval will be provided.

A regression model for censored data (Cox model) will explore prognostic factors. The IGIV immunological and pathological related efficacy endpoints will also be compared according to their distribution and analyzed using Student, Mann-Whitney and Fisher tests.

Other variables will be presented as means and standard deviations or medians and interquartile ranges according to their distribution and analyzed by Student, Mann-Whitney and Fisher tests.

Parameters that are measured on a time scale from randomization or start of administration will be compared between treatment groups using the Log-Rank test.

The choice of statistical tests and multivariate models (parametric or non-parametric) will be made for each variable based on observed characteristics (normality of distributions and residuals, collinearity).

The statistical analyses relating to the main objective will be carried out as intention to treat. Secondary analyses on the population per protocol may also be carried out.

All tests will be bilateral with a significance threshold of 5%. The software used will be SPSS v26 (SPSS Inc., Chicago, IL, USA). An interim analysis will be performed after 50 participants are enrolled and another after 100 inclusions.

ELIGIBILITY:
Inclusion Criteria:

* Any patient in intensive care:

  1. Receiving invasive mechanical ventilation for less than 72 hours
  2. ARDS meeting the Berlin criteria
  3. PCR-proven SARS-CoV-2 infection
  4. Patient, family or deferred consent (emergency clause)
  5. Affiliation to a social security scheme (or exemption from affiliation)

Exclusion Criteria:

* Allergy to polyvalent immunoglobulins
* Pregnant woman or minor patient
* Known IgA deficiency
* Patient with renal failure on admission defined by a 3 times baseline creatinine or creatinine >354 micromol/L or a diuresis of less than 0.3 mL/Kg for 24 hours or anuria for 12 hours
* Participation in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-04-11 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Ventilator-free days | 28 days
  Sum of the days the patient did not receive VM, but if death occurs before D28, the score is zero

SECONDARY OUTCOMES:
Mortality | 28 and 90 days
  Vital status at 28 and 90 days
Sequential Organ Failure Assessment Score | Days 1, 3, 7, 14, 21 and 28
  Used to determine the extent of a person's organ function or rate of failure, from 0 to 24, with severity increasing the higher the score
P/F ratio | Days 1, 3, 7, 14, 21 and 28
  Ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen (FiO2 expressed as a fraction, not a percentage)
Lung compliance | Days 1, 3, 7, 14, 21 and 28
  Measure of lung compliance
Radiological score | Days 1, 3, 7, 14, 21 and 28
  Severity scoring of lung oedema on the chest radiograph
Biological efficacy endpoints - C-reactive protein | Days 1, 3, 7, 14, 21 and 28
  Concentration in mg/L
Biological efficacy endpoints - Procalcitonin | Days 1, 3, 7, 14, 21 and 28
  Concentration in microgram/L
Immunological profile | Up to 28 days
  Number of CD4 HLA-DR+ and CD38+, CD8 lymphocytes
Number of patients using other treatments for COVID-19 related ARDS | Up to 28 days
  Use of corticosteroids, antiretroviral, chloroquine
Occurrence of deep vein thrombosis or pulmonary embolism | 28 days
  Diagnosis of deep vein thrombosis or pulmonary embolism through imaging exam (eg ultrasound and CT scan)
Total duration of mechanical ventilation, ventilatory weaning and curarisation | 28 days
  Total time of mechanical ventilation, weaning and use of neuromuscular blockade
Kidney Disease: Improving Global Outcomes (KDIGO) score and need for dialysis | 28 days
  Divided in 3 stages, with higher severity of kidney injury in higher stages
Occurrence of adverse event related to immunoglobulins | 28 days
  Kidney failure, hypersensitivity with cutaneous or hemodynamic manifestations, aseptic meningitis, hemolytic anemia, leuko-neutropenia, transfusion related acute lung injury (TRALI)
Occurrence of critical illness neuromyopathy | Up to 28 days
  Medical research council sum score on awakening
Occurrence of ventilator-acquired pneumonia | Up to 28 days
  Radiological and clinical context associated with a bacteriological sampling in culture of tracheal secretions, bronchiolar-alveolar lavage or a protected distal sampling

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Sharshar, MD, PHD, Study Chair — Centre Hospitalier Sainte Anne; Aurélien Mazeraud, MD, PHD, Principal Investigator — Centre Hospitalier Sainte Anne
Locations (42):
- France (42):
  - CHU Sud Amiens, Amiens
  - CHU Angers, Angers
  - Service de réanimation polyvalente, rond point de Girac, Angoulême
  - CH Victor Dupouy, Argenteuil
  - CH Aulnay, Aulnay-sous-Bois
  - Centre hospitalier de Béthune, Beuvry
  - Hopital Avicenne, Bobigny
  - CH-Nord-Ardennes, Charleville-Mézières
  - CH Chalons en champagne, Châlons-en-Champagne
  - Hopital d'instruction des armées Percy, Clamart
  - Centre Hospitalier de Dieppe, Dieppe
  - CH Etampes, Étampes
  - Hôpital Raymond Poincaré, Garches
  - CHU de Grenoble, Grenoble
  - Grand hopital de l'est Francilien - site de Jossigny, Jossigny
  - Hopital Robert Boulin, Libourne
  - Pôle de Médecine intensive/réanimation Hôpital Salengro, CHRU de Lille, Lille
  - Groupement Hospitalier Edouar Herriot, Lyon
  - Hôpital de la Croix Rousse Novembre 2019, Lyon
  - Hopital Jacques Cartier, Massy
  - Hopital Jacques Monod, Montivilliers
  - Service de Médecine Intensive-Réanimation, CHU, Nantes
  - CHR Orléans, Orléans
  - Centre Hospitalier Sainte-Anne, Paris
  - CHU Lariboisiere, Paris
  - CHU Pitié Salpétriere Service de réanimation chirurgicale, Paris
  - CHU Saint Antoine, Paris
  - Fondation ophtalmologique Rotschild, Paris
  - Hôpital Paris Saint-Joseph, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Poitiers, Poitiers
  - CHU Robert Débré, Reims
  - CH Poissy, Saint-Germain-en-Laye
  - Groupe hospitalier Saint Vincent, Strasbourg
  - Hôpital de Hautepierre, Strasbourg
  - Hopital de Tarbes, Tarbes
  - Hôpital Nord Franche-Comté, Trévenans
  - CH Valenciennes, Valenciennes
  - Chu Nancy - Brabois, Vandœuvre-lès-Nancy
  - Hopital de Vannes, Vannes
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Background] Chaigne B, Mouthon L. Mechanisms of action of intravenous immunoglobulin. Transfus Apher Sci. 2017 Feb;56(1):45-49. doi: 10.1016/j.transci.2016.12.017. Epub 2016 Dec 30. PMID 28161150
- [Background] Arish N, Eldor R, Fellig Y, Bogot N, Laxer U, Izhar U, Rokach A. Lymphocytic interstitial pneumonia associated with common variable immunodeficiency resolved with intravenous immunoglobulins. Thorax. 2006 Dec;61(12):1096-7. doi: 10.1136/thx.2004.029819. PMID 17114373
- [Background] Oates-Whitehead RM, Baumer JH, Haines L, Love S, Maconochie IK, Gupta A, Roman K, Dua JS, Flynn I. Intravenous immunoglobulin for the treatment of Kawasaki disease in children. Cochrane Database Syst Rev. 2003;2003(4):CD004000. doi: 10.1002/14651858.CD004000. PMID 14584002
- [Background] Alejandria MM, Lansang MA, Dans LF, Mantaring JB 3rd. Intravenous immunoglobulin for treating sepsis, severe sepsis and septic shock. Cochrane Database Syst Rev. 2013 Sep 16;2013(9):CD001090. doi: 10.1002/14651858.CD001090.pub2. PMID 24043371
- [Derived] Mazeraud A, Jamme M, Mancusi RL, Latroche C, Megarbane B, Siami S, Zarka J, Moneger G, Santoli F, Argaud L, Chillet P, Muller G, Bruel C, Asfar P, Beloncle F, Reignier J, Vinsonneau C, Schimpf C, Amour J, Goulenok C, Lemaitre C, Rohaut B, Mateu P, De Rudnicki S, Mourvillier B, Declercq PL, Schwebel C, Stoclin A, Garnier M, Madeux B, Gaudry S, Bailly K, Lamer C, Aegerter P, Rieu C, Sylla K, Lucas B, Sharshar T. Intravenous immunoglobulins in patients with COVID-19-associated moderate-to-severe acute respiratory distress syndrome (ICAR): multicentre, double-blind, placebo-controlled, phase 3 trial. Lancet Respir Med. 2022 Feb;10(2):158-166. doi: 10.1016/S2213-2600(21)00440-9. Epub 2021 Nov 11. PMID 34774185
- [Derived] Mazeraud A, Goncalves B, Aegerter P, Mancusi L, Rieu C, Bozza F, Sylla K, Siami S, Sharshar T. Effect of early treatment with polyvalent immunoglobulin on acute respiratory distress syndrome associated with SARS-CoV-2 infections (ICAR trial): study protocol for a randomized controlled trial. Trials. 2021 Feb 28;22(1):170. doi: 10.1186/s13063-021-05118-7. PMID 33648563

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-10-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT04350580/SAP_000.pdf